CLINICAL TRIAL: NCT06643702
Title: Screening for Benign Paroxysmal Positional Vertigo in Primary Care Among Elderly Presenting With Dizziness, Imbalance, and Increased Tendency to Fall
Brief Title: Prevalence av BPPV Among Elderly in Primary Care
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Emilija Rackauskaite, Resident doctor in General medicine, Region Stockholm
Other Study IDs: SLSO 2024-2982; 2024-05079-01 (Other: Swedish Ethical Review Authority (Etikprövningsmyndigheten))
Record Dates: First submitted 2024-10-13; First posted 2024-10-16 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Benign Paroxysmal Positional Vertigo (BPPV)
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study aims to investigate whether positional tests should be routinely performed on all elderly patients (65 years and older) presenting to primary care with symptoms of acute, episodic, or chronic dizziness or vertigo, unsteadiness, imbalance, and/or an increased tendency to fall in the past 12 months. Study aims to investigate whether diagnostic maneuvers should be performed regardless of the presence of conventional positional vertigo presentation associated with classical cases of benign paroxysmal positional vertigo (BPPV). Specifically, the study aims to identify "hidden" cases of BPPV and assess the potential benefits of clinical screening and initial treatment of BPPV in primary care setting thus improving the BPPV-related quality of life and reducing the risk of falls in the elderly population.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 65 years or older and present to the primary care clinic with one or several of the following:

1. Acute, episodic, or chronic sensation of dizziness/vertigo.
2. Subjective or objective imbalance during stance or movements.
3. Presented with increased tendency of falls by exhibiting unintentional loss of balance resulting in a fall one or more times in the past 12 months.

Exclusion Criteria:

1. Patients not meeting the above epidemiological and medical criteria described under "Inclusion Criteria".
2. Patients presenting with pathologies in which head and neck movements/manipulations are contraindicated, including (but not limited to): cervical instability, acute head and neck trauma, known cervical disk prolapse, Arnold-Chiari malformation, vascular pathologies such as carotid sinus syncope, vascular dissection and vertebrobasilarinsufficiency, including patients with paralysis as well as those with reduced mobility, in whom diagnostic maneuvers cannot be correctly performed.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Eligible participants are elderly patients aged 65 years and older who present to the primary care clinic with acute, episodic, or chronic dizziness or vertigo, unsteadiness, imbalance, and/or an increased tendency to fall by exhibiting unintentional loss of balance resulting in a fall one or more times in the past 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
What is the overall prevalence of BPPV among elderly patients (65 years and older) presenting with symptoms of dizziness, vertigo, unsteadiness, imbalance, or an increased tendency to fall in primary care setting? | From enrollment to the follow-up visit 2 weeks later in BPPV positive cases (only one visit for negative cases).

SECONDARY OUTCOMES:
What is the prevalence of benign paroxysmal positional vertigo among elderly patients seeking primary care for dizziness, unsteadiness, balance problems and/or an increased tendency to fall but not reporting conventional BPPV symptoms? | From enrollment to the follow-up visit 2 weeks later in BPPV positive cases (only one visit for negative cases).
  Outcome aims to identify prevalence of so-called hidden cases of BPPV.
What is the prevalence of benign paroxysmal positional vertigo among elderly patients seeking primary care for clear and well defined positional vertigo associated with conventional BPPV presentation? | From enrollment to the follow-up visit 2 weeks later in BPPV positive cases (only one visit for negative cases).
  Outcome aims to identify prevalence of so-called classical cases of BPPV.
What are the differences in demographic, clinical and life-quality results between BPPV-positive and BPPV-negative groups? | From enrollment to the follow-up visit 2 weeks later in BPPV positive cases (only one visit for negative cases).
  This outcome aims to evaluate differences between the two following patient groups: patients who present with symptoms but have no BPPV and patients who test positive for BPPV. Metrics that are analysed are: demographic information; current and previous diseases; current medications; frailty; Downtown fall risk index; fall risk according to "World guidelines for falls prevention and management for older adults: a global initiative", DHI-scores, TUG-test results, Dix-Hallpike-test result. Above mentioned metrics are not analysed between each other, instead the analysis is done for each metric between the two patient groups.
What are the differences in clinical and life-quality outcomes between so-called "classical" BPPV-cases and "hidden" BPPV-cases before and after treatment? | From enrollment to the follow-up visit 2 weeks later in BPPV positive cases (only one visit for negative cases).
  This outcome aims to evaluate differences in following patient groups: patients who present with conventional BPPV-related symptoms and test positive for BPPV and patients who present with more diffuse symptoms and experience imbalance in during stance or movements or have fallen in the past year and do not report the conventional BPPV symptoms but test positive for BPPV.
  Metrics that are analysed are: demographic information; current and previous diseases; current medications; frailty; Downtown fall risk index; fall risk according to "World guidelines for falls prevention and management for older adults: a global initiative", DHI-scores upon first visit and follow-up visit, TUG-test results, Dix-Hallpike-test result upon upon first visit and follow-up visit; referral status. Above mentioned metrics are not analysed between each other, instead the analysis is done for each metric between the two mentioned patient groups.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Verrecchia, PhD, Study Director — Karolinska Institutet
Locations (1):
- Boo health center, Saltsjö-Boo, Stockholm County, Sweden